CLINICAL TRIAL: NCT04612374
Title: Exploring the Acceptability and Efficacy of a Transdiagnostic Treatment for Misophonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00106807
Record Dates: First submitted 2020-10-27; First posted 2020-11-03 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-02

CONDITIONS: Misophonia
Keywords: Misophonia; Treatment
MeSH Terms: conditions — misophonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase 1: Unified Protocol, 2 week baseline (Experimental): Participants in this arm will complete two weeks of baseline assessment (during which they will complete questionnaires but not start treatment) and then receive 16 sessions of the Unified Protocol (UP). The UP is an emotion-focused treatment designed to teach participants skills to help manage difficult experiences.
  Interventions: Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders
- Phase 1: Experimental: Unified Protocol, 4 week baseline (Experimental): Participants in this arm will complete four weeks of baseline assessment (during which they will complete questionnaires but not start treatment) and then receive 16 sessions of the Unified Protocol (UP). The UP is an emotion-focused treatment designed to teach participants skills to help manage difficult experiences.
  Interventions: Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders
- Phase 2: Revised Unified Protocol, 2 week baseline (Experimental): Participants in this arm will complete two weeks of baseline assessment (during which they will complete questionnaires but not start treatment) and then receive 16 sessions of the revised Unified Protocol (UP). The UP is an emotion-focused treatment designed to teach participants skills to help manage difficult experiences and will be revised based on patient feedback in Phase 1.
  Interventions: Behavioral: Revised Unified Protocol for Transdiagnostic Treatment of Emotional Disorders
- Phase 2: Revised Unified Protocol, 4 week baseline (Experimental): Participants in this arm will complete four weeks of baseline assessment (during which they will complete questionnaires but not start treatment) and then receive 16 sessions of the revised Unified Protocol (UP). The UP is an emotion-focused treatment designed to teach participants skills to help manage difficult experiences and will be revised based on patient feedback in Phase 1.
  Interventions: Behavioral: Revised Unified Protocol for Transdiagnostic Treatment of Emotional Disorders

INTERVENTIONS:
Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders — Please see arm/group descriptions
  Arms: Phase 1: Experimental: Unified Protocol, 4 week baseline; Phase 1: Unified Protocol, 2 week baseline
Behavioral: Revised Unified Protocol for Transdiagnostic Treatment of Emotional Disorders — Please see arm/group descriptions
  Arms: Phase 2: Revised Unified Protocol, 2 week baseline; Phase 2: Revised Unified Protocol, 4 week baseline

SUMMARY:
Despite increasing recognition of misophonia, there are currently no evidence-based treatments to help those who are suffering. Therefore, the primary purpose of this study is to assess the acceptability, feasibility, and preliminary efficacy of a treatment for misophonia. This study will be conducted in two phases. In the Phase 1, participants will receive a treatment the investigators believe can help manage symptoms of misophonia: The Unified Protocol. This treatment uses evidence-based psychological principles (e.g., managing attention or behavior) in a flexible manner and will focus on developing skills to help reduce the distress and impairment associated with Misophonia. After treatment, patients will provide feedback about their experience. The investigators will use this feedback to revise the treatment as indicated. In Phase 2, participants will receive the revised treatment and provide feedback on their experience. Throughout treatment in either phase, participants will provide daily and weekly information about their symptoms.

The aims of this study are (1) to explore the acceptability and feasibility of the Unified Protocol for individuals who experience Misophonia and (2) to examine whether this treatment helps reduce symptoms associated with Misophonia.

ELIGIBILITY:
Inclusion Criteria:

* Between age 18-65
* Able to read English
* Meet criteria for interfering symptoms of misophonia
* Live in North Carolina

Exclusion Criteria:

* Under age 18 or over age 65
* Current mania
* Current psychotic disorder
* Current anorexia
* Presents with a condition that requires immediate prioritization in treatment (e.g., suicide planning or intent)

Phase 1 participants cannot also participate in Phase 2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
Number of patients that are satisfied with treatment as measured by the credibility and expectancy questionnaire (CEQ | up to 20 weeks
  The CEQ is a 6-item measure that asks patients about their perceptions of treatment.
Number of patients who indicate treatment was acceptable to them (i.e., the treatment approach made sense and was perceived as reasonable) | up to 20 weeks
  The Satisfaction with Therapy and Therapist Scale is a 13-item measure that asks patients about their satisfaction with treatment and with their therapist.
Number of sessions attended | up to 20 weeks
  The number of sessions attended will provide an estimate of the feasibility of attending and completing this treatment
Number of patients who use mindfulness skills assessed by the Southampton Mindfulness Questionnaire (SMQ) | up to 24 weeks
  The SMQ is a 16-item measure that asks patients about their use of mindfulness skills .
Number of patients who use cognitive flexibility skills assessed by the UP Cognitive Skills Questionnaire (CSQ) | up to 24 weeks
  The CSQ is a 10-item measure that assesses use of cognitive skills taught in treatment
Number of Patients who use behavior change skills assessed by the UP Behavioral Avoidance Questionnaire (BAQ) | up to 24 weeks
  The BAQ is a five item measure that assesses use of behavior change skills taught in treatment.
Number of patients who report a decrease in anxiety sensitivity on the Anxiety Sensitivity Index (ASI) | up to 24 weeks
  The ASI is an 18 measure that assesses how often a participant experiences anxiety symptoms
Number of Patients who use behavior change skills assessed by the Brief Experiential Avoidance Questionnaire (BEAQ) | up to 24 weeks
  The BEAQ is a 13 item measure that assesses how often a participant avoids emotion-provoking situations
Change in misophonia symptoms as assessed by the Misophonia Questionnaire | assessed weekly, up to 24 weeks
  The Misophonia Questionnaire is a 17-item questionnaire that assesses the presence of misophonia symptoms, emotions and behaviors associated with misophonic reactions, and symptom severity. The first two subscales are rated on a scale of 0 (not at all true) to 4 (always true). These two parts are summed to produce a total score ranging from 0 - 68. The severity subscale is a single item that asks an individual to provide a rating of their sound sensitivity on a scale from 0 (no sound sensitivities) to 15 (very severe sound sensitivities).
Change in anxiety as measured by the Overall Anxiety Severity and Impairment Scale | assessed weekly, up to 24 weeks
  The Overall Anxiety Severity and Impairment Scale is a five item measure that assesses interference and distress related to the experience of anxiety. Items are scored from 0 to 4 and summed to produce a total score (ranging from 0 - 20), with higher scores indicating greater functional impairment.
Change in depression as measured by the Overall Depression Severity and Impairment Scale | assessed weekly, up to 24 weeks
  The Overall Depression Severity and Impairment Scale is a five item measure that assesses interference and distress in an individual's day-to-day life related to the experience of depression. Items are scored from 0 to 4 and summed to produce a total score (ranging from 0 - 20), with higher scores indicating greater functional impairment.
Change in anger as measured by the PANAS Hostility Scale | assessed weekly, up to 24 weeks
  The PANAS Hostility Scale is a 6 item scale that assesses how often a participant experienced anger in the past week.

SECONDARY OUTCOMES:
Number of patients who report a change in attentional control as measured by the Digit Span Test | up to 20 weeks
  This test assesses a participant's ability to selectively use their attention during a task
Number of patients who report a change in attentional control as measured by the Trail Making Test | up to 20 weeks
  This test assesses a participant's ability to selectively use their attention during a task
Number of patients who report a change in cognitive flexibility as measured by the Stroop test | up to 20 weeks
  This test assesses a participant's ability to alternate their responses based on instructions.
Number of patients who report a change in cognitive flexibility as measured by the Trail Making Test | up to 20 weeks
  This test assesses a participant's ability to alternate their responses based on instructions.
Number of seconds participant engaged in a physiological challenge exercise | up to 20 weeks
  Participants will be asked to breathe through a small straw, with the option to stop at any time
Number of seconds participant engaged in a writing task | up to 20 weeks
  Participants will be asked to write about emotion-provoking situations, with the option to stop at any time

CONTACTS AND LOCATIONS:
Overall Officials: M. Zachary Rosenthal, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No